CLINICAL TRIAL: NCT03783949
Title: A Multicentre, Open-label, Three-arm Randomised Phase II Trial Assessing the Safety and Efficacy of the HSP90 Inhibitor Ganetespib in Combination With Carboplatin Followed by Maintenance Treatment With Niraparib Versus Ganetespib Plus Carboplatin Followed by Ganetespib and Niraparib Versus Carboplatin in Combination With Standard Chemotherapy Followed by Niraparib Maintenance Treatment in Platinum-sensitive Ovarian Cancer Patients
Brief Title: European Trial on Enhanced DNA Repair Inhibition in Ovarian Cancer
Acronym: EUDARIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-004058-40
Record Dates: First submitted 2018-12-14; First posted 2018-12-21 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Ganetespib; Niraparib
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — STA 9090; niraparib; Carboplatin; Paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Standard arm (arm A): Carboplatin (AUC5 d1, q3w i.v.) in combination with Paclitaxel (175 mg/m² d1, q3w i.v.) or Carboplatin (AUC4 d1, q3w i.v.) in combination with Gemcitabine (1000 mg/m² d1, d8, q3w i.v.) followed by maintenance therapy with Niraparib (200/ 300 mg oral daily, q4w) First experimental arm (arm B): Ganetespib (150 mg/m2, d1, q3w) in combination with Carboplatin (AUC5 d1, q3w i.v.) followed by maintenance treatment with Niraparib (200/ 300 mg oral daily, q4w) Second experimental arm (arm C): Ganetespib (150 mg/m² d1, q3w i.v.) plus Carboplatin (AUC5 d1, q3w i.v.) followed by Ganetespib (100 mg/m² d1, d8, d15, d22, q4w i.v.) and Niraparib (200 mg oral daily, q4w)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard arm (arm A) (Active Comparator): Carboplatin (AUC5 d1, q3w i.v.) in combination with Paclitaxel (175 mg/m² d1, q3w i.v.) or Carboplatin (AUC4 d1, q3w i.v.) in combination with Gemcitabine (1000 mg/m² d1, d8, q3w i.v.) followed by maintenance therapy with Niraparib (200/ 300 mg oral daily, q4w)
  Interventions: Drug: Niraparib; Drug: Carboplatin; Drug: Paclitaxel; Drug: Gemcitabine
- First experimental arm (arm B) (Experimental): Ganetespib (150 mg/m2, d1, q3w) in combination with Carboplatin (AUC5 d1, q3w i.v.) followed by maintenance treatment with Niraparib (200/ 300 mg oral daily, q4w)
  Interventions: Drug: Ganetespib; Drug: Niraparib; Drug: Carboplatin
- Second experimental arm (arm C) (Experimental): Ganetespib (150 mg/m² d1, q3w i.v.) plus Carboplatin (AUC5 d1, q3w i.v.) followed by Ganetespib (100 mg/m² d1, d8, d15, d22, q4w i.v.) and Niraparib (200 mg oral daily, q4w)
  Interventions: Drug: Ganetespib; Drug: Niraparib; Drug: Carboplatin

INTERVENTIONS:
Drug: Ganetespib — Ganetespib dose during chemotherapy will be 150mg/m² (q3w) Ganetespib dose during maintenance treatment will be 100mg/m² (q1w)
  Arms: First experimental arm (arm B); Second experimental arm (arm C)
Drug: Niraparib — Niraparib starting dose during maintenance treatment will be 200mg or 300mg depending on subject's body weight and subject neutrophil count (QD)
Drug: Carboplatin — In combination with Gemcitabine: Carboplatin dose will be AUC4 (q3w) In combination with Paclitaxel: Carboplatin dose will be AUC5 (q3w)
Drug: Paclitaxel — Paclitaxel dose will be 175mg/m² (q3w)
  Arms: Standard arm (arm A)
Drug: Gemcitabine — Gemcitabine dose will be 1000mg/m² (q3w, d1 & d8)
  Arms: Standard arm (arm A)

SUMMARY:
This study will be performed in women with platinum-sensitive, high-grade serous, high-grade endometrioid, undifferentiated epithelial ovarian cancer, carcinosarcoma, fallopian tube or primary peritoneal cancer (proven by central histo-pathological review).

A total of 120 subjects will be randomized (1:1:1) to three different treatment arms: (A) Standard arm (arm A): Carboplatin (AUC5 d1, q3w i.v.) in combination with Paclitaxel (175 mg/m² d1, q3w i.v.) or Carboplatin (AUC4 d1, q3w i.v.) in combination with Gemcitabine (1000 mg/m² d1, d8, q3w i.v.) followed by maintenance therapy with Niraparib (200/ 300 mg oral daily, q4w) // (B) First experimental arm (arm B): Ganetespib (150 mg/m2, d1, q3w) in combination with Carboplatin (AUC5 d1, q3w i.v.) followed by maintenance treatment with Niraparib (200/ 300 mg oral daily, q4w) // (C) Second experimental arm (arm C): Ganetespib (150 mg/m² d1, q3w i.v.) plus Carboplatin (AUC5 d1, q3w i.v.) followed by Ganetespib (100 mg/m² d1, d8, d15, d22, q4w i.v.) and Niraparib (200 mg oral daily, q4w).

Chemotherapy treatment will be given for 6 cycles, maintenance treatment with Ganetespib will be given for a maximum of 9 months or until disease progression, maintenance treatment with Niraparib can continue until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria to be eligible for study entry:

  * Ability to understand and willingness to sign and date a written informed consent document
  * Female patients ≥18 years of age
  * High-grade serous, high-grade endometrioid, undifferentiated epithelial ovarian cancer, carcinosarcoma, fallopian tube or primary peritoneal cancer
  * Platinum-sensitive relapse >6months after previous platinum-based treatment (calculated from the first day of the last cycle of the last platinum-based chemotherapy until the date of progression confirmed according to RECIST 1.1 on imaging)
  * No limits in number of prior lines
  * Measurable or evaluable disease according to RECIST 1.1
  * ECOG performance status 0-1
  * Adequate functions of the bone marrow
* Platelets ≥ 100 x 109/L
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L

  • Adequate function of the organs
* Creatinine < 2 mg/dl (<177 μmol/L)
* Total bilirubin ≤ 1.5 x upper limit of normal (≤ 2.0 in patients with known Gilberts syndrome) OR direct bilirubin ≤ 1 x ULN
* SGOT/SGPT (AST/ALT) ≤ 2.5 x upper limit of normal unless liver metastases are present, in which case they must be ≤ 5 x ULN
* Urinanalysis or urine dipstick for proteinuria less than 2+. Patients with ≥ 2+ on dipstick should undergo 24-hour urine collection and must demonstrate < 1 g of protein/24 hours; except the proteinuria is clearly related to a catheter in the urinary system.

  * Adequate coagulation parameter: aPTT ≤ 1.5 x ULN (patients on heparin treatment must have an aPTT between 1.5-2.5 x ULN), or INR ≤ 1.5. (In patients receiving anticoagulants (such as warfarin) INR must be between 2.0 and 3.0 in two consecutive measurements 1-4 days apart).
  * Participant receiving corticosteroids (dose < 10 mg/day methylprednisolone equivalent), including inhaled steroids, may continue as long as their dose is stable for at least 4 weeks prior to initiating protocol therapy.
  * Participants must agree to not donate blood during the study or for 90 days after the last dose of study treatment
  * Female participant has a negative serum pregnancy test within 7 days prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of non-childbearing potential. Non-childbearing potential is defined as follows (by other than medical reasons):
* ≥ 45 years of age and has not had menses for >1 year
* Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
* Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by imaging. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. See below for a list of acceptable birth control methods. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Birth Control: Participants of childbearing potential who are sexually active and their partners must agree to the use of a highly effective form of contraception throughout their participation beginning with time of consent, during the study treatment and for 180 days after last dose of study treatment(s):

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

    * Oral route
    * Intravaginal route
    * Transdermal route
  * Progestogen-only hormonal contraception associated with inhibition of ovulation

    * Oral
    * Injectable
    * Implantable
  * Intrauterine device
  * Intrauterine hormone-releasing system
  * Bilateral tubal occlusion
  * Vasectomized partner
  * Sexual abstinence, if the preferred and usual lifestyle of the subject

    * Participant must agree to not breastfeed (or store breast milk for use) during the study or for 180 days afer the last dose of study treatment.
    * Haemoglobin ≥8.5 g/dl (patients may not receive a transfusion within 4 weeks prior to initiating study treatment)
    * Able to take oral medications
    * Availability of archival ovarian cancer tissue from primary diagnosis (delivery of FFPE block or slides is prerequisite for randomisation)

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:

  * Ovarian tumours with low malignant potential (i.e. borderline tumours)
  * Any prior radiotherapy to the pelvis or abdomen, or any radiotherapy encompassing > 20 % of the bone marrow within 2 weeks, or any radiotherapy within 1 week prior to Day 1 of protocol therapy
  * Surgery (including open biopsy and traumatic injury) within 4 weeks prior to first dose of Ganetespib, or anticipation of the need for major surgery during study treatment
  * Minor surgical procedures, within 24 hours prior to the first study treatment
  * Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).

Any serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, chronic obstructive pulmonary disease, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.

* Current or recent (within 10 days prior to the first study drug dose) chronic daily treatment with aspirin (>325 mg/day).
* Patients with a history of diagnosis, detection or treatment of any prior malignancies ≤ 2 years prior to initiating protocol therapy, except: basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated.
* Clinically significant gastro-intestinal (GI) tract abnormalities that may increase the risk for GI bleeding and / or perforation including but not limited to: active peptic ulcer disease, known intraluminal metastatic lesion/s with risk of bleeding; inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), history of bowel obstruction within 1 year prior to first study treatment (excluding postoperative, i.e. within 4 weeks post surgery), other GI condition with increased risk of perforation such as recurrence deeply infiltrating into the muscularis or mucosa of the rectosigmoid or the mucosa of the bladder, or history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess
* Non-healing wound or non-healing bone fracture
* Patients with symptomatic brain or leptomeningeal metastases (patients who are asymptomatic since treatment of brain or leptomeningeal metastases, eg. after irradiation, are eligible)
* Left ventricular ejection fraction (LVEF) defined by ECHO below the institutional lower limit of normal
* Cerebrovascular accident (CVA)/ stroke or transient ischemic attack (TIA) or sub-arachnoid haemorrhage within ≤ 6 months prior to first study treatment.
* Significant cardiac disease: New York Heart Association (NYHA) Class 3 or 4; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty or coronary atrial or ventricular cardiac arrhythmias
* History of prolonged QT syndrome, or family member with prolonged QT syndrome
* QTc interval > 470 msec when 3 consecutive ECG values are averaged
* Ventricular tachycardia or a supraventricular tachycardia that requires treatment with a Class Ia antiarrhythmic drug (e.g. sotalol, amiodarone, dofetilide). Use of other antiarrhythmic drugs is permitted
* Second- or third-degree atrioventricular (AV) block, except: treated with a permanent pacemaker Complete left bundle branch block (LBBB)
* History of evidence of haemorrhagic disorders, patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorders, coagulopathy or tumour involving major vessels.
* Participation in another clinical study with experimental therapy within 28 days before start of treatment.
* Participant must not be simultaneously enrolled in any interventional clinical trial.
* Women who are pregnant or are lactating
* Patients unable to be regularly followed for any reason (geographic, familiar, social, psychologic, housed in an institution eg. prison because of a court agreement or administrative order)
* Subjects that are dependent on the sponsor/CRO or investigational site as well as on the investigator.
* History of known hypersensibility against any medication used in the study
* Intolerance / Hypersensitivity reactions to components and excipients of study drugs
* Peripheral neuropathy of grade >2 per NCI CTCAE, version 4.03, within 4 weeks prior to randomisation
* Any other condition that, in the opinion of the investigator, may compromise the safety, compliance of the patient, or would preclude the patient from successful completion of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 122 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- Medical University of Innsbruck, Innsbruck, Austria
- UZLeuven, Leuven, Vlaams-Brabant, Belgium
- France (3):
  - Centre de lutte contre le cancer Francois Baclesse, Caen
  - Centre anticancereux Leon Berard, Lyon
  - Assistance Publique Hôpitaux de Paris, Paris
- Germany (5):
  - Universitätsmedizin Berlin Charité, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Dresden, Dresden
  - Kliniken Essen Mitte, Evang. Huyssens- Stiftung/Knappschaft GmbH, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Italy (3):
  - Azienda Ospedaliero Bologna, Bologna
  - Fondazione IRCCS Istituto Nazionale dei tumori Milano, Milan
  - Università Cattolica del Sacro Cuore, Rome

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Arm (Arm A) | First Experimental Arm (Arm B) | Second Experimental Arm (Arm C)
Started | 41 | 42 | 39
Completed | 2 | 0 | 2
Not Completed | 39 | 42 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Arm (Arm A) | First Experimental Arm (Arm B) | Second Experimental Arm (Arm C) | Total
Number analyzed (Participants) | 41 | 42 | 39 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 25 | 22 | 68
  >=65 years | 20 | 17 | 17 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.77 (9.617) | 61.78 (13.097) | 62.76 (11.231) | 62.76 (11.357)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 39 | 122
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 41 | 42 | 39 | 122
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 2 | 1 | 4
  Belgium | 12 | 9 | 12 | 33
  Italy | 17 | 17 | 17 | 51
  France | 6 | 8 | 3 | 17
  Germany | 5 | 6 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 3 years 10 months
Population: The primary aim of this study was to determine the efficacy of the new agent regarding progression-free survival (PFS). Therefore the main analysis, as foreseen in the protocol, combined the two study arms with Ganetespib (arms B and C) and compare it against the standard arm (arm A).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Experimental Arms (Arm B&C): Ganetespib (150 mg/m2, d1, q3w) in combination with Carboplatin (AUC5 d1, q3w i.v.) followed by maintenance treatment:
  Arm B: Niraparib (200/ 300 mg oral daily, q4w) Arm C: Ganetespib (100 mg/m² d1, d8, d15, d22, q4w i.v.) and Niraparib (200 mg oral daily, q4w)
  Ganetespib: Ganetespib dose during chemotherapy will be 150mg/m² (q3w) Ganetespib dose during maintenance treatment will be 100mg/m² (q1w)
  Niraparib: Niraparib starting dose during maintenance treatment will be 200mg or 300mg depending on subject's body weight and subject neutrophil count (QD)
  Carboplatin: In combination with Gemcitabine: Carboplatin dose will be AUC4 (q3w) In combination with Paclitaxel: Carboplatin dose will be AUC5 (q3w)
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 41 | 80
months | 8.85 [7.73 to 11.55] | 8.32 [6.88 to 9.70]

2. Secondary Outcome: Progression-free Survival in BRCA Mutated Patients
Description: Progression-free survival analysis in BRCA mutated patients
Time Frame: 3 years 10 months
Population: The primary aim of this study was to determine the efficacy of the new agent regarding progression-free survival (PFS). Therefore the main analysis, as foreseen in the protocol, combined the two study arms with Ganetespib (arms B and C) and compare it against the standard arm (arm A), both for the primary outcome as for all secondary and exploratory outcomes.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 13 | 24
months | 11.78 [7.30 to 17.37] | 7.98 [6.09 to 11.05]

3. Secondary Outcome: Post-progression PFS (PFS2)
Description: Post-progression PFS (PFS2) analysis
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 41 | 79
months | 21.71 [17.73 to 25.30] | 21.38 [15.53 to 26.18]

4. Secondary Outcome: Time to First Subsequent Therapy (TFST)
Description: Time to First Subsequent Therapy (TFST) analysis
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 41 | 80
months | 9.38 [8.09 to 12.47] | 8.75 [7.40 to 10.07]

5. Secondary Outcome: Time to Second Subsequent Therapy (TSST)
Description: Time to Second Subsequent Therapy (TSST) analysis
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 41 | 80
months | 17.73 [14.28 to 21.61] | 14.54 [13.26 to 16.94]

6. Secondary Outcome: Progression-free Survival in Patients Without BRCA Mutation or With Unknown BRCA Status
Description: Progression-free Survival analysis in Patients without BRCA mutation or with unknown BRCA status
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 28 | 56
months | 7.83 [6.58 to 11.38] | 8.49 [6.71 to 10.49]

7. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) analysis
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Standard Arm (Arm A): Carboplatin (AUC5 [AUC=Area under the curve] d1, q3w i.v. [q3w=every three weeks, i.v.=intravenously]) in combination with Paclitaxel (175 mg/m² d1, q3w i.v. [q3w=every three weeks, i.v.=intravenously]) or Carboplatin (AUC4 [AUC=Area under the curve] d1, q3w i.v. [q3w=every three weeks, i.v.=intravenously]) in combination with Gemcitabine (1000 mg/m² d1, d8, q3w i.v. [q3w=every three weeks, i.v.=intravenously]) followed by maintenance therapy with Niraparib (200/ 300 mg oral daily, q4w [q4w=every four weeks])
  Niraparib: Niraparib starting dose during maintenance treatment will be 200mg or 300mg depending on subject's body weight and subject neutrophil count (QD) [QD=once daily].
  Carboplatin: In combination with Gemcitabine: Carboplatin dose will be AUC4 (q3w) [AUC=area under the curve, q3w=every three weeks] In combination with Paclitaxel: Carboplatin dose will be AUC5 (q3w) [AUC=area under the curve, q3w=every three weeks]
  Paclitaxel: Paclitaxel dose will be 175mg/m² (q3w) [q3w=every three weeks]
  Gemcitabine: Gemcitabine dose will be 1000mg/m² (q3w, d1 & d8) [q3w=every three weeks]
- Experimental Arms (Arm B&C): Ganetespib (150 mg/m2, d1, q3w [q3w=every three weeks]) in combination with Carboplatin (AUC5 [AUC=Area under the curve] d1, q3w i.v. [q3w=every three weeks, i.v.=intravenously]) followed by maintenance treatment:
  Arm B: Niraparib (200/ 300 mg oral daily, q4w [q4w=every four weeks]) Arm C: Ganetespib (100 mg/m² d1, d8, d15, d22, q4w i.v. [q4w=every four weeks, i.v.=intravenously])) and Niraparib (200 mg oral daily, q4w [q4w=every four weeks])
  Ganetespib: Ganetespib dose during chemotherapy will be 150mg/m² (q3w [q3w=every three weeks]) Ganetespib dose during maintenance treatment will be 100mg/m² (q1w [q1w=every week])
  Niraparib: Niraparib starting dose during maintenance treatment will be 200mg or 300mg depending on subject's body weight and subject neutrophil count (QD) [QD=once daily].
  Carboplatin: In combination with Gemcitabine: Carboplatin dose will be AUC4 (q3w) [q3w=every three weeks] In combination with Paclitaxel: Carboplatin dose will be AUC5 (q3w) [q3w=every three weeks]
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 38 | 79
Participants
  no response (SD/PD) | 21 | 52
  response (PR/CR) | 17 | 27

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) analysis
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 41 | 81
months | 22.14 [17.73 to 29.97] | 22.27 [17.07 to 29.21]

9. Secondary Outcome: Progression-free Survival in Patients With Prior PARPi Treatment
Description: Progression-free Survival analysis in Patients with prior PARPi treatment
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 13 | 25
months | 7.40 [5.63 to 8.85] | 6.09 [2.76 to 7.76]

10. Secondary Outcome: Progression-free Survival in Patients With One Prior Line of Therapy
Description: Progression-free Survival analysis in Patients with one prior line of therapy
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 27 | 46
months | 10.59 [5.92 to 11.94] | 9.70 [7.14 to 11.35]

11. Secondary Outcome: Progression-free Survival in Patients With More Then One Prior Line of Therapy
Description: Progression-free Survival analysis in Patients with more then one prior line of therapy
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 14 | 34
months | 7.63 [7.30 to 12.89] | 7.43 [4.11 to 8.32]

12. Secondary Outcome: Progression-free Survival in Patients Without Prior PARPi Treatment
Description: Progression-free Survival analysis in Patients without prior PARPi treatment
Time Frame: 3 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard Arm (Arm A) | Experimental Arms (Arm B&C)
Number analyzed (Participants) | 28 | 55
months | 11.55 [7.43 to 13.55] | 9.77 [7.83 to 11.12]

ADVERSE EVENTS:
Time Frame: 3 years 10 months
Description: This trial consisted of a first period in which chemotherapy (CT) was administered and of a maintenance treatment (MT) period. Not all patients completed the CT or were allowed to start in the MT. Both groups were analyzed separately in order to differentiate between CT and MTevents. This result section does not accommodate for the separate reporting both groups so we reported all events in this section, differentiation can be made based on the number of patients that were at risk.
Groups:
- Standard Arm (Arm A) - Chemotherapy Phase: Carboplatin (AUC5 d1, q3w i.v.) in combination with Paclitaxel (175 mg/m² d1, q3w i.v.) or Carboplatin (AUC4 d1, q3w i.v.) in combination with Gemcitabine (1000 mg/m² d1, d8, q3w i.v.) followed by maintenance therapy with Niraparib (200/ 300 mg oral daily, q4w)
  Niraparib: Niraparib starting dose during maintenance treatment will be 200mg or 300mg depending on subject's body weight and subject neutrophil count (QD)
  Carboplatin: In combination with Gemcitabine: Carboplatin dose will be AUC4 (q3w) In combination with Paclitaxel: Carboplatin dose will be AUC5 (q3w)
  Paclitaxel: Paclitaxel dose will be 175mg/m² (q3w)
  Gemcitabine: Gemcitabine dose will be 1000mg/m² (q3w, d1 & d8)
- First Experimental Arm (Arm B) - Chemotherapy Phase: Ganetespib (150 mg/m2, d1, q3w) in combination with Carboplatin (AUC5 d1, q3w i.v.) followed by maintenance treatment with Niraparib (200/ 300 mg oral daily, q4w)
  Ganetespib: Ganetespib dose during chemotherapy will be 150mg/m² (q3w) Ganetespib dose during maintenance treatment will be 100mg/m² (q1w)
  Niraparib: Niraparib starting dose during maintenance treatment will be 200mg or 300mg depending on subject's body weight and subject neutrophil count (QD)
  Carboplatin: In combination with Gemcitabine: Carboplatin dose will be AUC4 (q3w) In combination with Paclitaxel: Carboplatin dose will be AUC5 (q3w)
- Second Experimental Arm (Arm C) - Chemotherapy Phase: Ganetespib (150 mg/m² d1, q3w i.v.) plus Carboplatin (AUC5 d1, q3w i.v.) followed by Ganetespib (100 mg/m² d1, d8, d15, d22, q4w i.v.) and Niraparib (200 mg oral daily, q4w)
  Ganetespib: Ganetespib dose during chemotherapy will be 150mg/m² (q3w) Ganetespib dose during maintenance treatment will be 100mg/m² (q1w)
  Niraparib: Niraparib starting dose during maintenance treatment will be 200mg or 300mg depending on subject's body weight and subject neutrophil count (QD)
  Carboplatin: In combination with Gemcitabine: Carboplatin dose will be AUC4 (q3w) In combination with Paclitaxel: Carboplatin dose will be AUC5 (q3w)
- Standard Arm (Arm A) - Maintenance Phase: Carboplatin (AUC5 d1, q3w i.v.) in combination with Paclitaxel (175 mg/m² d1, q3w i.v.) or Carboplatin (AUC4 d1, q3w i.v.) in combination with Gemcitabine (1000 mg/m² d1, d8, q3w i.v.) followed by maintenance therapy with Niraparib (200/ 300 mg oral daily, q4w)
  Niraparib: Niraparib starting dose during maintenance treatment will be 200mg or 300mg depending on subject's body weight and subject neutrophil count (QD)
- First Experimental Arm (Arm B) - Maintenance Phase: Ganetespib (150 mg/m2, d1, q3w) in combination with Carboplatin (AUC5 d1, q3w i.v.) followed by maintenance treatment with Niraparib (200/ 300 mg oral daily, q4w)
  Ganetespib: Ganetespib dose during chemotherapy will be 150mg/m² (q3w)
- Second Experimental Arm (Arm C) - Maintenance Phase: Ganetespib (150 mg/m² d1, q3w i.v.) plus Carboplatin (AUC5 d1, q3w i.v.) followed by Ganetespib (100 mg/m² d1, d8, d15, d22, q4w i.v.) and Niraparib (200 mg oral daily, q4w)
  Ganetespib: Ganetespib dose during chemotherapy will be 150mg/m² (q3w)
Arm/Group | Standard Arm (Arm A) - Chemotherapy Phase | First Experimental Arm (Arm B) - Chemotherapy Phase | Second Experimental Arm (Arm C) - Chemotherapy Phase | Standard Arm (Arm A) - Maintenance Phase | First Experimental Arm (Arm B) - Maintenance Phase | Second Experimental Arm (Arm C) - Maintenance Phase
All-Cause Mortality (participants affected / at risk) | 41/41 | 42/42 | 39/39 | 32/32 | 26/26 | 17/17
Serious Adverse Events (participants affected / at risk) | 20/41 | 19/42 | 16/39 | 13/32 | 8/26 | 5/17
Other Adverse Events (participants affected / at risk) | 40/41 | 42/42 | 39/39 | 32/32 | 26/26 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Arm (Arm A) - Chemotherapy Phase (N=41) | First Experimental Arm (Arm B) - Chemotherapy Phase (N=42) | Second Experimental Arm (Arm C) - Chemotherapy Phase (N=39) | Standard Arm (Arm A) - Maintenance Phase (N=32) | First Experimental Arm (Arm B) - Maintenance Phase (N=26) | Second Experimental Arm (Arm C) - Maintenance Phase (N=17)
CRP increased (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (General disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
allergic reaction NOS (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction to Carboplatin (Immune system disorders) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ascites (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fistula (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
general deterioration (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal subobstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney insufficiency (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maligne pleuritis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Investigations) | 8 (8) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Tumor biopsy (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastro-entiritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Word finding disorders (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Arm (Arm A) - Chemotherapy Phase (N=41) | First Experimental Arm (Arm B) - Chemotherapy Phase (N=42) | Second Experimental Arm (Arm C) - Chemotherapy Phase (N=39) | Standard Arm (Arm A) - Maintenance Phase (N=32) | First Experimental Arm (Arm B) - Maintenance Phase (N=26) | Second Experimental Arm (Arm C) - Maintenance Phase (N=17)
QTc prolongation (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
abdominal cramping (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (General disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction to Carboplatin (Immune system disorders) | 6 (6) | 9 (9) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Alopecia (General disorders) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Investigations) | 32 (32) | 26 (26) | 25 (25) | 18 (18) | 12 (12) | 7 (22)
Anorexia (General disorders) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Asthenia (General disorders) | 12 (12) | 16 (16) | 10 (10) | 2 (2) | 4 (4) | 6 (16)
blurry vision (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (11) | 7 (7) | 9 (9) | 7 (7) | 5 (5) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 19 (19) | 20 (20) | 3 (3) | 3 (3) | 12 (40)
Dizziness (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 10 (10) | 7 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
General malaise (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (General disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 6 (6) | 3 (3)
Insomnia (General disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Leucocytopenia (Investigations) | 28 (28) | 12 (12) | 10 (10) | 10 (10) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (22) | 25 (25) | 16 (16) | 10 (10) | 7 (7) | 13 (13)
Neutropenia (Investigations) | 35 (55) | 19 (26) | 17 (22) | 0 (0) | 0 (0) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1) | 17 (17) | 6 (6) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Syncope (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Investigations) | 35 (35) | 29 (29) | 29 (29) | 11 (11) | 14 (14) | 5 (5)
Transaminases increased (Investigations) | 11 (11) | 5 (5) | 6 (6) | 3 (3) | 2 (2) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (6) | 11 (11) | 9 (9) | 3 (3) | 4 (4) | 7 (7)
QTcF prolongation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal bloating (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alkaline phosphatase increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dysgeusia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 5 (5)
Hypertension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
itching (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
Weight decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT03783949/Prot_SAP_000.pdf